CLINICAL TRIAL: NCT05101122
Title: Open-Label 4-Period Dose-Escalation Safety and Efficacy Study of AD313 in Participants With Obstructive Sleep Apnea
Brief Title: Study for Efficacy and Dose Escalation of AD313 + Atomoxetine (SEED)
Acronym: SEED
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SEED
Record Dates: First submitted 2021-10-07; First posted 2021-11-01 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Apnea, Obstructive Sleep; Sleep Apnea Syndromes; Upper Airway Reistance Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dosing Period 1: Atomoxetine (Active Comparator): 3 days of atomoxetine 40 mg followed by 4 days of atomoxetine 80 mg.
  Interventions: Drug: Dosing 1: Atomoxetine
- Dosing Period 2-4: AD313 (Experimental): Week 2: atomoxetine 40 mg/dronabinol 2.5 mg Week 3: atomoxetine 80 mg/dronabinol 5 mg Week 4: atomoxetine 80 mg/dronabinol 10 mg
  Interventions: Drug: AD313

INTERVENTIONS:
Drug: Dosing 1: Atomoxetine — Oral administration at bedtime
  Other Names: 40mg or 80 mg Atomoxetine
  Arms: Dosing Period 1: Atomoxetine
Drug: AD313 — Escalating dose of AD313; Oral administration at bedtime
  Other Names: atomoxetine dronabinol
  Arms: Dosing Period 2-4: AD313

SUMMARY:
The SEED study is designed to assess the safety and efficacy for Obstructive Sleep Apnea (OSA) of 3 escalating dose combinations of atomoxetine with AD313 compared to baseline and to atomoxetine alone.

DETAILED DESCRIPTION:
The SEED study is an open-label, 4 consecutive period dose-escalation study of combinations of AD313 vs. atomoxetine alone in participants with moderate- to severe OSA. A screening polysomnogram (PSG) will be conducted to establish that each participant meets study enrollment criteria and to serve as baseline. Each participant will then receive escalating doses of AD313 with on-drug PSGs to be conducted on the final night of dosing.

ELIGIBILITY:
Inclusion Criteria:

Age and Sex

1. 25 to 65 years of age, inclusive, at the Screening Visit. Disease Measures
2. AHI 10 to 50 (hypopneas defined by 4% oxygen desaturation)
3. ≤25% of apneas are central or mixed apneas at V2 baseline PSG Weight
4. BMI between 18.5 and 40.0 kg/m2, inclusive, at the pre-PSG visit.

   Male participants:
5. If male and sexually active with female partner(s) of childbearing potential, participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (see Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information).

   Female participants:
6. If a woman of childbearing potential (WOCBP), the participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (See Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information). All WOCBP must have negative result of a serum pregnancy test performed at screening.
7. If female and of non-childbearing potential, the participant must be either postmenopausal (defined as age ≥ 55 years with no menses for 12 or more months without an alternative medical cause) or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

   Informed Consent
8. Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening Visit procedures.
9. Participant must be able to understand the nature of the study and must have the opportunity to have any questions answered.

Exclusion Criteria:

Medical Conditions

1. History of clinically significant sleep disorder other than OSA.
2. Clinically significant craniofacial malformation.
3. Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control (combination medications are considered as 1 medication for this purpose).
4. Clinically significant neurological disorder, including epilepsy/convulsions.
5. History of schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM 5) or International Classification of Disease tenth edition criteria.
6. History of attempted suicide within 1 year prior to screening, or current suicidal ideation.
7. Medically unexplained positive screen for drugs of abuse or history of substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.
8. A significant illness or infection requiring medical treatment in the past 30 days.
9. Clinically significant cognitive dysfunction as determined by investigator.
10. Women who are pregnant or nursing. Prior/Concomitant Therapy
11. History of using devices for OSA treatment, including CPAP, oral or nasal devices, or positional devices, may enroll as long as the devices have not been used for at least 2 weeks prior to first study visit and are not used during participation in the study.
12. History of chronic oxygen therapy.
13. Use of medications from the list of disallowed concomitant medications.
14. Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, strong cytochrome P450 2D6 (CYP2D6) inhibitors, or monoamine oxidase inhibitors (MAOI) within 14 days of the start of treatment, or concomitant with treatment.

    Prior/Concurrent Clinical Study Experience
15. Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.

    Diagnostic Assessments
16. Hepatic transaminases >2X the upper limit of normal (ULN), total bilirubin >1.5X ULN (unless confirmed Gilbert syndrome), estimated glomerular filtration rate < 60 ml/min.
17. PLM arousal index >15 Other Exclusions
18. <5 hours typical sleep duration.
19. ESS > 18
20. Night- or shift-work sleep schedule which causes the major sleep period to be during the day.
21. Employment as a commercial driver or operator of heavy or hazardous equipment.
22. Typically smoking more than 10 cigarettes or 2 cigars per day, or inability to abstain from smoking during overnight PSG visits.
23. Unwilling to use specified contraception.
24. History of regular alcohol consumption of more than 14 standard units per week (males) or more than 7 standard units per week (females), or unwillingness to limit alcohol consumption to no greater than 2 units/day (males), 1 unit per day (females), not to be consumed within 3 hours of bedtime or on PSG nights.
25. Unwilling to limit during the study period caffeinated beverage intake (e.g., coffee, cola, tea) to 400 mg/day or less of caffeine, not to be used within 3 hours of bedtime.
26. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.
27. Participant considered by the investigator, for any reason, an unsuitable candidate to receive atomoxetine and/or dronabinol or unable or unlikely to understand or comply with the dosing schedule or study evaluations.

Meals and Dietary Restrictions

1. Participants should refrain from consumption of any nutrients known to modulate CYP enzyme activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, pomegranate, and Seville or Moro [blood] orange products) within 72 hours before the first dose of study drug and during the study.
2. Diet should be generally stable during the study, e.g., new diet programs should not be initiated.

Caffeine, Alcohol, and Tobacco

1. During the outpatient portions of the study, participants should refrain from more than 2 standard units per day of alcohol for men or 1 unit/day for women, consumed no less than 3 hours prior to bedtime. Alcohol should not be consumed on PSG nights.
2. Moderate consumption of caffeinated beverages, containing up to a total of 400 mg caffeine per day, is permitted during the study period, consumed no less than 3 hours prior to bedtime.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Farkas, MD, PhD, Study Director — Apnimed Inc.
Locations (2):
- United States (2):
  - Santa Monica Clinical Trials, Los Angeles, California
  - Clayton Sleep Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messineo L, Norman D, Ojile J. The combination of atomoxetine and dronabinol for the treatment of obstructive sleep apnea: a dose-escalating, open-label trial. J Clin Sleep Med. 2023 Jul 1;19(7):1183-1190. doi: 10.5664/jcsm.10528. PMID 36805833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited from an existing medical clinic and will have up to three weeks screening.
Groups:
- Dosing Periods: Participants who meet all enrollment criteria will receive an escalating dose of atomoxetine the first week: 3 days of atomoxetine 40 mg followed by 4 days of atomoxetine 80 mg. Participants will then receive escalating dose combinations of atomoxetine and dronabinol for the next 3 weeks.
Period: Atomoxetine Only
Arm/Group | Dosing Periods
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: AD313 40/2.5
Arm/Group | Dosing Periods
Started | 14
Completed | 12
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: AD313 80/5
Arm/Group | Dosing Periods
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: AD313 80/10
Arm/Group | Dosing Periods
Started | 11
Completed | 10
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: This analysis was performed according to a modified intention-to-treat procedure, namely after inclusion of all participants who took at least one dose of any study medication and had at least one efficacy measure
Arm/Group | Dosing Periods
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Body Mass Index (BMI) [Median (Standard Deviation); unit: kg/m2] | 31.9 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI)4% Events Per Hour
Description: Compares high dose atomoxetine (80/10) versus baseline
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: events/hour
Groups:
- Baseline: Participants at baseline
- AD313 80/10: Atomoxetine 80 mg/ dronabinol 10 mg
Arm/Group | Baseline | AD313 80/10
Number analyzed (Participants) | 15 | 10
events/hour | 28.6 [16.19 to 33.65] | 26.6 [8.78 to 31.93]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 9 weeks
Groups:
- Dosing Period 1: Atomoxetine Alone; Dosing Period 3: Atomoxetine 40 + Dronabinol 2.5 mg; Dosing Period 4: Atomoxetine 80 + Dronabinol 5mg; Dosing Period 5: Atomoxetine 80 + Dronabinol 10mg: Participants who meet all enrollment criteria received an escalating dose of atomoxetine the first week: 3 days of atomoxetine 40 mg followed by 4 days of atomoxetine 80 mg. Participants then received escalating dose combinations of atomoxetine and dronabinol for the next 3 weeks.
Arm/Group | Dosing Period 1: Atomoxetine Alone | Dosing Period 3: Atomoxetine 40 + Dronabinol 2.5 mg | Dosing Period 4: Atomoxetine 80 + Dronabinol 5mg | Dosing Period 5: Atomoxetine 80 + Dronabinol 10mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 9/15 | 7/14 | 6/12 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dosing Period 1: Atomoxetine Alone (N=15) | Dosing Period 3: Atomoxetine 40 + Dronabinol 2.5 mg (N=14) | Dosing Period 4: Atomoxetine 80 + Dronabinol 5mg (N=12) | Dosing Period 5: Atomoxetine 80 + Dronabinol 10mg (N=11)
Hypersomnia (Nervous system disorders) | 2 | 0 | 1 | 0
Impotence, erectile dysfunction (Reproductive system and breast disorders) | 3 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dizziness, lightheadedness (Nervous system disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vasomotor symptoms - Hot flashes (Vascular disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Jitteriness (Nervous system disorders) | 1 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Night time sweating (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Paranoia (Psychiatric disorders) | 0 | 1 | 1 | 0
Paresthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 — Subject withdrew during period 3 because started having suicidal thoughts and no longer wanted to continue.
Tingling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — The morning after he takes study medication, he has a constant tingling feeling on his head/hair and it lasts all day.
Dissociative state (Psychiatric disorders) | 0 | 0 | 0 | 1 — Subject reported feeling dissociated from her body 30 mins after dosing IP- resolved by the time she went to sleep.
Urinary hesitancy (Renal and urinary disorders) | 2 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Xerostomia (Gastrointestinal disorders) | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

The Sponsor retains the right to disapprove any submission for publication, including any publication using trial data, including abstracts, presentations or manuscripts.

A summary of the study results will also be posted in a publicly accessible database (e.g., www.ClinTrials.gov).

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT05101122/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT05101122/ICF_001.pdf